CLINICAL TRIAL: NCT03946826
Title: A Clinical Observation on the Efficacy and Safety of Pulsed Dye Laser (PDL) in the Treatment of Nail Psoriasis: a Single-blind, Randomized, Self-controlled Trial
Brief Title: A Clinical Observation on the Efficacy and Safety of Pulsed Dye Laser (PDL) in the Treatment of Nail Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: xjpfW (Other)
Collaborators: Air Force General Hospital of the PLA (Other Government); First Hospital of China Medical University (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, xjpfW, Head of Dermatology, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: XJPFMR-20150707
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Nail Psoriasis
Keywords: nail psoriasis; Pulsed dye laser (PDL); Halometasone Cream; Vaseline
MeSH Terms: interventions — Petrolatum; Lasers, Dye

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PDL+ Halometasone Cream group (Experimental): PDL+ Halometasone Cream Halometasone Cream, bid ,external use for 6 months; 3 nails were randomly selected to be treated with PDL laser therapy (6ms, 11±2J/cm2) once a month for a total of 6 times
  Interventions: Drug: Halometasone Cream; Radiation: Pulsed dye laser (PDL)
- PDL+Vaseline group (Experimental): PDL+Vaseline Vaseline, bid ,external use for 6 months; 3 nails were randomly selected to be treated with PDL laser therapy (6ms, 11±2J/cm2) once a month for a total of 6 times
  Interventions: Drug: Vaseline; Radiation: Pulsed dye laser (PDL)
- Halometasone Cream (Active Comparator): Halometasone is a potent halogen - containing topical glucocorticoid. Have stronger fight inflammation, fight allergy, contractive hemal, reduce hemal to connect the action of permeability and fight hyperplasia
  Interventions: Drug: Halometasone Cream
- Vaseline (Placebo Comparator): Vaseline belongs to a kind of mineral wax, without irritant, not easy to deteriorate, can let skin surface form a protective film when used on the skin, let the moisture of the skin be evaporated not easily, have better protect wet effect
  Interventions: Drug: Vaseline

INTERVENTIONS:
Drug: Halometasone Cream — Halometasone is a potent halogen - containing topical glucocorticoid. Have stronger fight inflammation, fight allergy, contractive hemal, reduce hemal to connect the action of permeability and fight hyperplasia
  Arms: Halometasone Cream; PDL+ Halometasone Cream group
Drug: Vaseline — Vaseline belongs to a kind of mineral wax, without irritant, not easy to deteriorate, can let skin surface form a protective film when used on the skin, let the moisture of the skin be evaporated not easily, have better protect wet effect
  Arms: PDL+Vaseline group; Vaseline
Radiation: Pulsed dye laser (PDL) — Pulsed dye laser (PDL) is effective for vasodilatory diseases, especially for the superficial to middle layers of the dermis,is effective in the treatment of psoriasis
  Arms: PDL+ Halometasone Cream group; PDL+Vaseline group

SUMMARY:
1. Psoriasis is a common chronic, inflammatory disease characterized by skin changes and joint involvement. About 50% of patients with psoriasis have damage to the nail, especially in pustular psoriasis in the continuous acromegaly dermatitis. Common damage includes pitting, uneven and tarnish of the deck, as well as the occurrence of nail ridges, furrows, turbidity, hypertrophy, free ends and nail bed stripping, and even the whole deck deformity or absence, etc., seriously affecting patients' social interaction and mental health. Pathologically, telangiectasis is associated with the superficial and middle layers of the dermis. Previous treatment of psoriasis nail is mainly topical drugs (such as glucocorticoid, etc.), but due to its long disease period, topical drugs are difficult to transdermal absorption, and the curative effect of skin lesions is poor.
2. Pulsed dye laser (PDL) is effective for vasodilatory diseases, especially for the superficial to middle layers of the dermis
3. It has been reported that PDL is effective in the treatment of psoriasis vulgis by blocking the nutrient supply vessels of the lesions, improving the surrounding microenvironment, reducing the number of cytotoxic T cells and helper T cells in the dermis, and promoting the normalization of epidermal proliferation and differentiation.
4. Halometasone is a potent halogen - containing topical glucocorticoid. Have stronger fight inflammation, fight allergy, contractive hemal, reduce hemal to connect the action of permeability and fight hyperplasia Vaseline belongs to a kind of mineral wax, without irritant, not easy to deteriorate, can let skin surface form a protective film when used on the skin, let the moisture of the skin be evaporated not easily, have better protect wet effect.

ELIGIBILITY:
Inclusion Criteria:

.subjects must be clinically diagnosed by the investigator to have nail psoriasis .All nails have psoriasis on both hand.Males or females, 18 Years to 65 Years of age at the time of signing the informed consent document.

.No other external treatment was performed before the injury was treated. .The condition of no rupture or infection in the skin affected the field of vision of laser operation.

.The patient has no history of treatment of biological preparations, such as Indolisimab, etc.

.Check blood routine, liver and kidney function, normal blood sugar, female urine pregnancy test negative during childbearing age.

.Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.

Exclusion Criteria:

* Pregnant or lactating women with a history of light sensitivity;
* The patient has just stopped or started new systemic treatment; Patients with serious infectious diseases;
* suffering from severe diabetes, severe cardiovascular disease and connective tissue disease;
* patients with a history of active tuberculosis, blood diseases, and epilepsy;
* There are infected persons and patients with acute infectious diseases in the treatment site;
* Patients who are considered by the researchers to be unfit to participate in this experiment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
NAPSI score | Change from Baseline to 1 year
  1. Nail matrix score: according to the proportion of nail matrix damage (puncture, meniscus with all white and red spots, and nail fragmentation) to the nail matrix content, 0 means no, 1 means 1/4 nail, 2 means 2/4 nail, 3 means cumulative 3/4 nail, and 4 means total nail.
  2. Nail bed score: the nail bed damage (nail dissection, puncture hemorrhage, hyperkeratosis under the nail, salmon spot) is graded according to the proportion of the nail bed. 0 means no, 1 means 1/4 nail, 2 means 2/4 nail, 3 means cumulative 3/4 nail, and 4 means total nail.
  3. Single nail score is the sum of nail matrix score and nail bed score (0-8 points), The final score is the sum of all single nail scores (0-80), and the nail score can be conducted at any time as required.

SECONDARY OUTCOMES:
VAS Pain Assessment | Change from Baseline to 6 months
  VAS Pain Assessment，Immediately after Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wang Gang, Prof, Principal Investigator — Dermatology Derpartment of Xijing Hospital

IPD SHARING:
Plan to Share IPD: No